CLINICAL TRIAL: NCT04804189
Title: Reframing Firearm Injury Prevention Through Bystander Interventions for Youth Shooting Sports Participants
Brief Title: Reframing Firearm Injury Prevention Through Bystander Interventions for Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Nicole Nugent, Psychologist, Rhode Island Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01CE003267 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-03-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-08

CONDITIONS: Firearm Injury
Keywords: firearm injury prevention; bystander intervention; youth violence prevention; shooting sports; firearm safety

STUDY DESIGN:
Intervention Model Description: We will enroll up to 60 4-H Shooting Sports communities nationwide to participate in a Type I Hybrid Effectiveness Trial. All Clubs will receive standard national-level training and curricula. Clubs randomized to "Guardians 4 Health" intervention will add additional training to enable Club Leaders to integrate Guardians 4 Health methods into their standard activities. We will provide ongoing technical support to all intervention Clubs. In all enrolled communities, we will measure 1) short- and intermediate-term outcomes among both Club-level adult and teen leaders and the Club's youth participants and their primary caregivers, and 2) injury incidence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Up to 30 4-H Shooting Sport Clubs that will not receive Guardians 4 Health intervention.
- Intervention Group (Experimental): Up to 30 Randomized 4-H Shooting Sport Clubs that will receive Guardians 4 Health intervention.
  Interventions: Behavioral: Guardians 4 Health

INTERVENTIONS:
Behavioral: Guardians 4 Health — Clubs will implement Guardians 4 Health's intervention into their community by incorporating Guardians 4 Health materials into standard Club educational activities.
  Arms: Intervention Group

SUMMARY:
Modifiable risk factors for youth firearm injury and death include unsafe storage of a firearm in the home, prior victimization/aggression, substance use, and depressive symptoms, yet there are few partnerships with firearm owners and firearm safety training programs to implement effective, non-policy-based preventive interventions for youth firearm injury. This study will conduct a hybrid effectiveness-implementation trial to evaluate the effectiveness of Guardians 4 Health, a bystander intervention designed to promote changes in firearm injury prevention norms, attitudes, intentions, and behaviors among a sample up to 60 4-H Shooting Sports Club communities comprising both adults and youth. This project is designed to build the evidence base for interventions that promote safe behaviors related to youth firearm use and injury prevention and advance firearm injury prevention science by supporting a synergistic partnership between well-established firearm injury, suicide, and violence prevention researchers and the national 4-H Shooting Sports community.

DETAILED DESCRIPTION:
Firearm injury and mortality is a major public health concern for American youth age 1-19. Only motor vehicle crashes kill more American youth than firearms. In 2018 alone, 1729 American youth died from firearm injuries (50% firearm homicide, 42% firearm suicide) and over 6500 youth were treated in an emergency department for firearm injury; these injuries have major long-term consequences for youth and their families. Approximately one-third of American youth live in a home with a firearm. Risk factors for youth firearm injury and death, such as unsafe home storage of a firearm, prior victimization/aggression, substance use, and depressive symptoms, can be modified. Community partnerships are essential for developing and enacting effective change in injury risk factors, particularly for youth. Due to the fraught political landscape and lack of research funding, partnerships with firearm owners and firearm safety training programs to create and disseminate effective, non-policy-based preventive interventions for youth firearm injury are lacking.

Bystander intervention (BI) is an intervention framework rooted in social psychological theories such as the Theory of Planned Behavior (TPB), with proven efficacy and effectiveness targeting both individual and community behavior change. "Guardians 4 Health" is a three-part, already-piloted intervention that uses the BI framework and TPB mechanisms to promote community norms change about firearm safety, BI, and harm reduction techniques (e.g., safe storage, reducing access to lethal means, conflict resolution). Recognizing that BI is most rigorous when led by credible messengers, Guardians 4 Health uses instructional, peer-to-peer, and social-media strategies in conjunction with community organizations that are deeply connected to firearm safety efforts. Pilot data supports Guardian 4 Health's acceptability and feasibility in changing firearm owners' norms and behaviors.

The necessary next step in this intervention development is to evaluate its effectiveness using a randomized, controlled study design. Our community partner, the National 4-H Shooting Sports Program, is a national leader and trusted messenger for firearm safety. Across the United States, 20,000 trained adult Club Leaders, 5,000 Teen Ambassadors, and 450,000 youth Shooting Sports participants (age 8-18) learn marksmanship, and safe and responsible use of firearms, through its structured curriculum. Leaders from 4-H are excited to implement and study Guardian 4 Health among their Shooting Sports Clubs and communities to reduce youth firearm injury and mortality risk. Our research team will evaluate Guardian 4 Health's effectiveness, compared to usual 4-H training, in changing firearm injury prevention norms, attitudes, behavioral intention, and practice among a sample of one hundred 4-H Shooting Sports Club communities, via a Type I Hybrid randomized, controlled effectiveness trial. Aims are:

Refinement and Planning (Year 1): Adapt Guardians 4 Health for the 4-H Shooting Sports Club context Aim 1: Conduct a series of key informant interviews with an advisory panel of up to 40 key stakeholders (teen and adult 4-H Shooting Sports leaders representing a diverse group of communities and 4-H experience) to ensure The Reframe addresses 4-H-specific issues of acceptability, feasibility, and appropriateness.

Intervention Delivery (Years 2-3): Conduct a hybrid Type I effectiveness-implementation trial of Guardians 4 Health with up to 60 4-H Shooting Sports communities across the United States. For each intervention site, we will engage one Adult Site Champion in a kickoff meeting; provide materials to incorporate into standard 4-H curricula; and provide ongoing technical support. Evaluations will be conducted at 0, 3, and 6 months.

Aim 2A: Evaluate Guardian 4 Health's effectiveness, compared to usual training, in changing individual- and community-level, proximal and distal behavioral outcomes related to firearm injury prevention.

Aim 2B: Examine barriers and facilitators to implementation of Guardians 4 Health intervention using a mixed-methods (qualitative and quantitative) approach.

Aim 2C: (Exploratory) Explore injury patterns among all participating communities using population-level data.

The study will advance the science of firearm injury prevention in youth in the context of a real-world partnership between well-established firearm injury, suicide, and violence prevention researchers and the National 4-H Shooting Sports Program to conduct a rigorous experimental evaluation of a promising universal primary prevention program. Our long-term goals, consistent with CDC priorities, are to build an evidence base for best practices for individual- and community-level interventions that are easy to implement; to promote safe behaviors around firearm use and injury prevention, thereby saving lives; to meld best scientific practice with deep community-based expertise; and to create a model that can be scaled across 4-H's network, which reaches nearly 6 million youth across the nation.

ELIGIBILITY:
Inclusion Criteria:

* Membership of child participant in local 4-H Shooting Sports Club OR
* Parent of a child participant in local 4-H Shooting Sports Club OR
* Community member of a participating local 4-H Shooting Sports Club

Exclusion Criteria:

* Non-English speakers
* Unable to consent or assent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Change in Intention to Use Behavioral Intervention Skills via Cook-Craig et al 2014 | 0, 3 and 6 months
  We will measure intention to intervene to prevent firearm injury using a scale adapted from Cook-Craig et al 2014.
  Scale title: Adapted Theory of Planned Behavior Scale Minimum value: 1 Maximum value: 5 Higher score (adjusted for reverse coding) indicates a better outcome.
  Due to under-enrollment, the study team decided to have this outcome as the SINGLE primary outcome in September 2024, before any data analysis began.

SECONDARY OUTCOMES:
Feasibility of Intervention via Percent of Intervention Activities Completed | 3 and 6 months
  We will use a target of 75% of participants completing intervention activities as a means of assessing intervention feasibility. Standard implementation metrics (e.g., on number of 4-H Club sessions, number of community events, number of participants at each Community event) will also be collected.
Change in Perceived Behavioral Control via Adapted Theory of Planned Behavior Scale | 0, 3 and 6 months
  Perceived behavioral control regarding intervention as a bystander will be measured using a scale adapted from Azjen's Theory of Planned Behavior (1).
  Scale title: Adapted Theory of Planned Behavior Scale Minimum value: 1 Maximum value: 5 Higher score (adjusted for reverse coding) indicates a better outcome.
Change in Subjective Norms via Adapted Theory of Planned Behavior Scale | 0, 3 and 6 months
  Norms regarding both firearm safety and bystander intervention will be measured using a scale adapted from Azjen's Theory of Planned Behavior (1).
  Scale title: Adapted Theory of Planned Behavior Scale Minimum value: 1 Maximum value: 5 Higher score (adjusted for reverse coding) indicates a better outcome.
Change in Attitudes via Adapted Theory of Planned Behavior Scale | 0, 3 and 6 months
  Attitudes regarding both firearm injury prevention and bystander intervention will be measured using a scale adapted from Azjen's Theory of Planned Behavior (Citation not indexed in PubMed: Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991;50(2):179-211.)
  Scale title: Adapted Theory of Planned Behavior Scale Minimum value: 1 Maximum value: 5 Higher score (adjusted for reverse coding) indicates a better outcome.
Change in Knowledge of Firearm Injuries in the US | 0, 3 and 6 months
  Knowledge of frequency, types, and risk factors for firearm injury will be assessed using a series of true/false questions based on intervention content.
Acceptability of Intervention via The Ottawa Acceptability Scale | 3 and 6 months
  The Ottawa Acceptability Scale (OAS) measures multiple dimensions of acceptability of an intervention including: length; amount of information; balance in presentation of information; and overall appropriateness for the community. The OAS is a 15-item scale (most with 4-point Likert scale response options) that will be assessed from all enrolled participants (Site Champions, Teen Ambassadors, Club Leaders, youth participants, and primary caregivers) at all time points. We will use a target of 85% of participants rating Guardians 4 Health as acceptable (global rating). Standard implementation metrics (e.g., on number of 4-H Club sessions, number of community events, number of participants at each Community event) will also be collected.
Barriers to Intervention via Qualitative Interviews Using the Consolidated Framework for Intervention Research | 3 and 6 months
  Measured qualitatively via semi-structured interviews with Site Champions and a purposefully sampled subset of adult Club Leaders, as guided by the Proctor Implementation Outcomes framework. These interviews will be structured using the Consolidated Framework for Intervention Research; we will query around barriers at the level of the intervention, outer setting (national 4-H, surrounding community), inner setting (local Club), and individual (adult leader) level.
Facilitators of Intervention via Qualitative Interviews Using the Consolidated Framework for Intervention Research | 3 and 6 months
  Measured qualitatively via semi-structured interviews with Site Champions and a purposefully sampled subset of adult Club Leaders, as guided by the Proctor Implementation Outcomes framework. These interviews will be structured using the Consolidated Framework for Intervention Research; we will query around barriers at the level of the intervention, outer setting (national 4-H, surrounding community), inner setting (local Club), and individual (adult leader) level.

OTHER OUTCOMES:
Change in Use of Behavioral Intervention Skills via Cook-Craig et al 2014 | 0, 3, and 6 months
  This measure will be adapted from a previously validated survey by Cook-Craig et al 2014.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Nugent, PhD, Principal Investigator — Brown University
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
We will provide an open dataset containing anonymized IPD that results in a publication, along with open code from our analyses, and open access to research articles. The PIs will document collected data using the Data Documentation Initiative (DDI), which is recommended by the national data archive: the Inter-university Consortium for Political and Social Research (ICPSR). Audio interviews of participants consenting to be recorded will be transcribed and de-identified; audio recordings will not be available for analysis due to concerns about re-identifiability. Transcripts will only be available with participant consent, and de-identified transcripts would be made available to other researchers via a Data Use Agreement (DUA) facilitated by ICPSR.
  We will deposit the aggregate data sets, survey and semi-structured interview instruments, analysis code, NVivo codes and associated codebook and relevant README documentation files in the ICPSR data archive.
Supporting Information: Analytic Code
Time Frame: Within 30 months of completing data collection.
Access Criteria: Data files deposited into ICPSR receive a Digital Object Identifier (DOI), which the Investigators will cite and include in all publications for the public and other researchers to locate and access the data. The Investigators will comply with the CDC Public Access Policy and upon acceptance deposit the final peer-reviewed manuscript of publications in PubMed Central (PMC), CDC Stacks, and Investigators' institutional repositories for free and public access.
URL: https://www.icpsr.umich.edu/web/pages/

REFERENCES:
- [Background] Cook-Craig PG, Coker AL, Clear ER, Garcia LS, Bush HM, Brancato CJ, Williams CM, Fisher BS. Challenge and opportunity in evaluating a diffusion-based active bystanding prevention program: Green Dot in high schools. Violence Against Women. 2014 Oct;20(10):1179-202. doi: 10.1177/1077801214551288. Epub 2014 Sep 24. PMID 25255794
- [Background] Ajzen I. The theory of planned behavior. Organizational Behavior and Human Decision Processes. 1991;50(2):179-211.
- [Result] Trinka T, Oesterle DW, Silverman AC, Vriniotis MG, Orchowski LM, Beidas RS, Betz ME, Hudson C, Kesner T, Ranney ML. Bystander intervention to prevent firearm injury: A qualitative study of 4-H shooting sports participants. J Community Psychol. 2023 Sep;51(7):2652-2666. doi: 10.1002/jcop.23069. Epub 2023 Jun 9. PMID 37294273